CLINICAL TRIAL: NCT06717334
Title: Enrichment of Lung Cancer Screening Through Unexplained Weight Loss (UWL) to Stage Shift and Improve Survival
Brief Title: A Study of Lung Cancer Screening in People With Unexplained Weight Loss
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-302
Record Dates: First submitted 2024-12-03; First posted 2024-12-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer Screening
Keywords: ctDNA analysis; Low dose computed tomography (CT)
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Lung cancer screening: All patients will undergo prospective LDCT imaging annually. At baseline and Year 1, patients will also undergo biospecimen collection for post-hoc ctDNA analysis.
  Interventions: Diagnostic Test: Low Dose CT imaging; Other: blood draws; Other: screening questionnaire

INTERVENTIONS:
Diagnostic Test: Low Dose CT imaging — at baseline and at Year 1.
Other: blood draws — at baseline and at Year 1.
Other: screening questionnaire — at baseline and at 1 year after registration.

SUMMARY:
The researchers are doing this study to see if people with unexplained weight loss who have lung cancer screening are more likely to have or develop lung cancer than people without unexplained weight loss. The lung cancer screening will involve use of low-dose computed tomography (LDCT), a CT scan that gives off very low doses of radiation and can make detailed pictures of the lungs to help find tumors. The study researchers will also analyze participants' blood samples to determine if blood testing can be used to help to diagnose lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for American Cancer Society lung cancer screening, as follows:

  * Age 50-80 years old
  * At least 20-pack year history of smoking
* Weight loss of 3-10%, defined as UWL, within any timeframe over the past in the 18 months prior to enrollment, that cannot be attributed to an underlying medical condition at the discretion of the enrolling investigator

  * Note that patients who have 3-10% weight may still be enrolled if the enrolling investigator does not conclude that the weight loss can be attributed to the patient's intentional efforts.
  * Documented weight loss can be self-reported or extracted from weights obtained during physician visits. However, if self-reported weight loss is contradicted by weight loss documented in the medical record (e.g. a patients states that (s)he lost 10 lbs in the past 6 months, but a weight documented in the medical record does not support that history), the measured and quantified weight change will be used to ascertain eligibility
* Life expectancy greater than 1 year, per assessment of the treating clinician.

Exclusion Criteria:

* Currently pregnant or trying to become pregnant via self-report
* Prior history of recent CT scan of the chest either through LDCT screening or with a scan of the chest (standard, not LDCT) performed within the past 12 months
* Prior history of NSCLC

  ○ Note that patients with a history of diagnosis of non-lung cancers are eligible for the study.
* Currently undergoing or referred for diagnostic evaluation due to clinical suspicion for malignancy (e.g., referred to a medical or surgical oncologist, or scheduled for biopsy on the basis of a suspicious imaging abnormality).
* Patients with a germline pathogenic genetic variant who have undergone whole body MRI within the past 12 months
* Unable to comply with study procedures

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified at MSKCC largely through survivorship clinics.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of lung cancer in patients with unexplained weight loss | 2 years
  Low Dose CT screening

CONTACTS AND LOCATIONS:
Overall Officials: Puneeth Iyengar, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Montefiore Health Systems (Montefiore Medical Center), The Bronx, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm